CLINICAL TRIAL: NCT03422718
Title: Reach Out: Randomized Clinical Trial of Emergency Department-Initiated Hypertension Behavioral Intervention Connecting Multiple Health Systems
Brief Title: Reach Out: Emergency Department-Initiated Hypertension Behavioral Intervention Connecting Multiple Health Systems
Acronym: ReachOut ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, William J Meurer, Associate Professor of Emergency Medicine, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HUM00138470; R01MD011516 (NIH)
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: stroke; hypertension
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1 (Experimental): No healthy behavior texts BP Monitoring Weekly Via Text Messaging No physician appointment and transportation scheduling
  Interventions: Behavioral: No healthy behavior texts; Behavioral: BP Monitoring Weekly Via Text Messaging; Behavioral: No physician appointment and transportation scheduling
- Arm 2 (Experimental): Healthy Behavior Texts BP Monitoring Weekly Via Text Messaging No physician appointment and transportation scheduling
  Interventions: Behavioral: Healthy Behavior Texts; Behavioral: BP Monitoring Weekly Via Text Messaging; Behavioral: No physician appointment and transportation scheduling
- Arm 3 (Experimental): No healthy behavior texts BP Monitoring Daily Via Text Messaging No physician appointment and transportation scheduling
  Interventions: Behavioral: No healthy behavior texts; Behavioral: BP Monitoring Daily Via Text Messaging; Behavioral: No physician appointment and transportation scheduling
- Arm 4 (Experimental): Healthy Behavior Texts BP Monitoring Daily Via Text Messaging No physician appointment and transportation scheduling
  Interventions: Behavioral: Healthy Behavior Texts; Behavioral: BP Monitoring Daily Via Text Messaging; Behavioral: No physician appointment and transportation scheduling
- Arm 5 (Experimental): No healthy behavior texts BP Monitoring Weekly Via Text Messaging Physician appointment and transportation scheduling
  Interventions: Behavioral: No healthy behavior texts; Behavioral: BP Monitoring Weekly Via Text Messaging; Behavioral: Physician appointment and transportation scheduling
- Arm 6 (Experimental): Healthy Behavior Texts BP Monitoring Weekly Via Text Messaging Physician appointment and transportation scheduling
  Interventions: Behavioral: Healthy Behavior Texts; Behavioral: BP Monitoring Weekly Via Text Messaging; Behavioral: Physician appointment and transportation scheduling
- Arm 7 (Experimental): No healthy behavior texts BP Monitoring Daily Via Text Messaging Physician appointment and transportation scheduling
  Interventions: Behavioral: No healthy behavior texts; Behavioral: BP Monitoring Daily Via Text Messaging; Behavioral: Physician appointment and transportation scheduling
- Arm 8 (Experimental): Healthy Behavior Texts BP Monitoring Daily Via Text Messaging Physician appointment and transportation scheduling
  Interventions: Behavioral: Healthy Behavior Texts; Behavioral: BP Monitoring Daily Via Text Messaging; Behavioral: Physician appointment and transportation scheduling

INTERVENTIONS:
Behavioral: Healthy Behavior Texts — Participants receive motivational health behavior texts
  Arms: Arm 2; Arm 4; Arm 6; Arm 8
Behavioral: No healthy behavior texts — Participants do not receive healthy behavior texts
  Arms: Arm 1; Arm 3; Arm 5; Arm 7
Behavioral: BP Monitoring Daily Via Text Messaging — Daily text messages will prompt participants for BP by home cuff
  Arms: Arm 3; Arm 4; Arm 7; Arm 8
Behavioral: BP Monitoring Weekly Via Text Messaging — Weekly text messages will prompt participants for BP by home cuff
  Arms: Arm 1; Arm 2; Arm 5; Arm 6
Behavioral: Physician appointment and transportation scheduling — Participants receive assistance scheduling physician appointment and transportation to those appointments
  Arms: Arm 5; Arm 6; Arm 7; Arm 8
Behavioral: No physician appointment and transportation scheduling — Participants do not receive assistance scheduling physician appointment or transportation
  Arms: Arm 1; Arm 2; Arm 3; Arm 4

SUMMARY:
This study evaluates a health theory based mobile health behavioral intervention to reduce blood pressure (BP) among hypertensive patients evaluated in a community Emergency Department (ED) setting.

DETAILED DESCRIPTION:
Hypertension is the most important modifiable risk factor for cardiovascular disease, the leading cause of mortality in the United States. African Americans have the highest prevalence of hypertension of any race/ethnic group in the United States which largely contributes to their increased burden of stroke compared to non-Hispanic whites. In addition, uncontrolled hypertension is more common among socioeconomically disadvantaged populations than their counterparts. To improve health equity, new approaches to hypertension treatment focusing on health care systems and difficult-to-reach populations are needed.

The Emergency Department (ED) represents a missed opportunity to identify and treat hypertension in difficult-to-reach populations. Currently, there are 136 million ED visits per year and nearly all have at least one blood pressure measured and recorded. African Americans and socioeconomically disadvantaged patients are disproportionally represented in the ED patient population and both are increasing. In the age of electronic health records and mobile health, the ED can feasibly become an integral partner in chronic disease management by programming the electronic health record to identify hypertensive patients and dispense a mobile health behavioral intervention. Facilitating ED follow up at primary care clinics is a key feature of the proposed intervention. Thereby leveraging the strengths of the ED and its large patient volume of uncontrolled, difficult-to-reach, hypertensive patients, with the strengths of the primary care clinics, continuity of care is the key to improving community wide utilization of health services and receipt of guideline concordant medical care.

This study looks to determine which behavioral intervention components best contribute to a reduction in systolic blood pressure at one year through a multi-component theory based mobile health behavioral intervention.

Sample Size and Population

We originally planned to enroll approximately 960 patients into the eligibility phase. From this group, we estimate that 480 participants will report qualifying BPs and will be randomized to one of the eight intervention arms. We anticipate 240 participants will fully complete the 12 month, in person follow up visits. However, after accruing approximately 400 randomized participants, we noted lower than expected retention at 6 month visits. Therefore, we adjusted the maximum total number of enrollments and randomizations upwards by 50% each. The overall intention is to achieve approximately 240 protocol completers (attendees at 12-month visit). We will continue to monitor accrual and retention in order to achieve this target.

Data Analysis

The primary analysis will fit a linear regression model with the outcome of SBP change (baseline minus 12 months) and main effect-coded binary predictors of healthy behavior texts (yes vs. no), prompted BP self-monitoring frequency (high vs. low), and primary care provider visit scheduling and transportation (active vs. passive). Initial analyses will focus on the main effects. Additional analyses will include all the two-way interactions of the three intervention components (only considering interactions where at least one of the factors in the interaction demonstrates a sufficiently large main effect).

The main secondary analyses will use time-to event (Cox Proportional Hazards) and logistic regression. For the endpoint of interest, (either time to first primary care visit, or the binary variable indicating attendance at two or more primary care visits within 1 year of randomization), the investigators will fit an adjusted regression model.

Extension Study:

Reach Out Cognition which will extend Reach Out data collection past the current 12 months to 15 and 18 months. During Reach Out Cognition, we aim to assess novel approaches to mobile health (mHealth) self-administered cognition and blood pressure (BP) measurements. These approaches may include cognitive assessments via mobile applications (apps) and Web-based surveys, and wireless BP measurements via Bluetooth-enabled blood pressure cuffs and apps.

The study population for Reach Out Cognition will be drawn from Reach Out participants who complete the Reach Out intervention and are defined as: participants who complete the 12-month outcome assessment. We anticipate about 240 participants will have completed Reach Out's 12-month outcome assessment and will be eligible for Reach Out Cognition.

Descriptive statistics will be used to evaluate acceptability, feasibility and satisfaction. The de-nominator is the number of Reach Out participants who complete the 12 month assessments. Regarding feasibility, we will separately determine the feasibility by mHealth measure (i.e. cognition vs. BP), phone type (i.e. smartphone vs. feature phone) and operating system type (iOS vs. Android vs. Windows) as a continuous and dichotomous (>50% completion of each assessment type) measure. The satisfaction scale will be assessed for all participants. Given the difference in procedures by phone type, we will compare satisfaction between the smartphone and feature phone users using a Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or greater
* At least one BP with Systolic Blood Pressure (SBP) ≥ 160 or a Diastolic Blood Pressure (DBP) ≥ 100 (criteria 1)
* If the patient has repeated measurements after achieving Criteria 1, at least one of the repeat BP remains SBP ≥ 140 or a DBP ≥ 90
* Must have cell phones with text-messaging capability and willingness to receive texts
* Likely to be discharged from the ED

Exclusion Criteria:

* Unable to read English (<1% at study site)
* Prisoners
* Pregnant
* Pre-existing condition making one year follow-up unlikely

  * Terminal illness with death expected within 90 days
* Current use of 3 or more antihypertensive agents
* Patients with other serious medical conditions that prevent self-monitoring of BP
* Critical illness with placement in resuscitation bay
* Dementia/cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Meurer, MD, Principal Investigator — University of Michigan; Lesli Skolarus, MD, Principal Investigator — University of Michigan; Mackenzie Dinh, MS, Study Director — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
In accordance with NIH policy, a public use dataset will be prepared by the investigators. The archiving and posting procedures are to be determined at this point.

REFERENCES:
- [Derived] Dinh M, Lin CC, Whitfield C, Farhan Z, Meurer WJ, Bailey S, Skolarus LE. Exploring the Acceptability and Feasibility of Remote Blood Pressure Measurements and Cognition Assessments Among Participants Recruited From a Safety-Net Emergency Department (Reach Out Cognition): Nonrandomized Mobile Health Trial. JMIR Form Res. 2024 May 28;8:e54010. doi: 10.2196/54010. PMID 38805251
- [Derived] Skolarus LE, Dinh M, Kidwell KM, Lin CC, Buis LR, Brown DL, Oteng R, Giacalone M, Warden K, Trimble DE, Whitfield C, Farhan Z, Flood A, Borgialli D, Montas S, Jaggi M, Meurer WJ. Reach Out Emergency Department: A Randomized Factorial Trial to Determine the Optimal Mobile Health Components to Reduce Blood Pressure. Circ Cardiovasc Qual Outcomes. 2023 May;16(5):e009606. doi: 10.1161/CIRCOUTCOMES.122.009606. Epub 2023 May 16. PMID 37192282
- [Derived] Skolarus LE, Dinh M, Kidwell KM, Farhan Z, Whitfield C, Levine DA, Meurer WJ. Supplement study update for Reach Out: a multi-arm randomized trial of behavioral interventions for hypertension initiated in the emergency department: Reach Out Cognition. Trials. 2021 Nov 24;22(1):836. doi: 10.1186/s13063-021-05806-4. PMID 34819115
- [Derived] Meurer WJ, Dinh M, Kidwell KM, Flood A, Champoux E, Whitfield C, Trimble D, Cowdery J, Borgialli D, Montas S, Cunningham R, Buis LR, Brown D, Skolarus L. Reach out behavioral intervention for hypertension initiated in the emergency department connecting multiple health systems: study protocol for a randomized control trial. Trials. 2020 Jun 3;21(1):456. doi: 10.1186/s13063-020-04340-z. PMID 32493502

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in Flint, Michigan, an urban, low-income, predominately Black community. Participants were recruited from the city's only safety-net ED (i.e., hospitals where over 25% of patients are Medicaid recipients). Enrollment occurred between March 2019 and March 2020.
Pre-assignment Details: Participants entered a run-in phase of 3 weeks to determine whether a participant had persistently elevated BP. During this time, participants were prompted to text their BP once per week to the study team. Participants responding at least once and with at least one systolic BP ≥ 140 or a diastolic BP ≥ 90 were randomized.
Period: 12 Month Interventional Trial Period
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Started | 62 | 60 | 63 | 61 | 58 | 61 | 64 | 59
6 Month Outcome | 26 | 35 | 30 | 29 | 31 | 32 | 29 | 28
Completed (Completed here means completed 12 month outcomes) | 25 | 31 | 25 | 22 | 30 | 31 | 24 | 23
Not Completed | 37 | 29 | 38 | 39 | 28 | 30 | 40 | 36
Not completed — Lost to Follow-up | 26 | 16 | 23 | 27 | 21 | 22 | 36 | 25
Not completed — Withdrawal by Subject | 11 | 13 | 15 | 12 | 7 | 8 | 4 | 11
Period: Optional Six Month Follow-Up Period
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Started (This simply represents all those who completed the 12 month and had the option to continue; some chose not to exercise it) | 25 | 31 | 25 | 22 | 30 | 31 | 24 | 23
Opted in to Optional Follow Up Phase (Note: Although participants are shown here based on the arm in which they participated during the main 12 month study, there was) | 17 | 20 | 9 | 8 | 13 | 17 | 10 | 13
Completed | 1 | 1 | 1 | 2 | 2 | 2 | 5 | 3
Not Completed | 24 | 30 | 24 | 20 | 28 | 29 | 19 | 20
Not completed — Chose Not to start 6 month extension | 8 | 11 | 16 | 14 | 17 | 14 | 14 | 10
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — ineligible | 8 | 5 | 2 | 2 | 1 | 5 | 2 | 4
Not completed — Lost to Follow-up | 8 | 11 | 6 | 4 | 9 | 8 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8 | Total
Number analyzed (Participants) | 62 | 60 | 63 | 61 | 58 | 61 | 64 | 59 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.6) | 47.7 (11.8) | 49 (11.4) | 45.3 (11.7) | 45.5 (12.5) | 46.5 (12.2) | 45.6 (12.6) | 45.3 (12.2) | 45.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 38 | 37 | 36 | 38 | 39 | 37 | 299
  Male | 25 | 23 | 25 | 24 | 22 | 23 | 25 | 22 | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 2 | 3 | 2 | 2 | 1 | 17
  Not Hispanic or Latino | 59 | 59 | 60 | 59 | 55 | 59 | 62 | 58 | 471
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 29 | 29 | 34 | 31 | 35 | 39 | 35 | 30 | 262
  White | 28 | 27 | 27 | 29 | 19 | 19 | 27 | 25 | 201
  More than one race | 5 | 2 | 1 | 1 | 4 | 3 | 2 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 60 | 63 | 61 | 58 | 61 | 64 | 59 | 488
Prior medication for hypertension within the last 6 months [Count of Participants; unit: Participants] | 35 | 35 | 34 | 34 | 33 | 33 | 36 | 33 | 273
Currently have a primary care provider [Count of Participants; unit: Participants] | 51 | 50 | 45 | 48 | 47 | 47 | 49 | 43 | 380

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Systolic Blood Pressure
Description: Change in 12-month Systolic Blood Pressure (SBP)
Time Frame: 12 months
Population: numbers analyzed in each row show all the participants at the two timepoints (baseline and 12 month) for which data exists.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8
Number analyzed (Participants) | 62 | 60 | 63 | 61 | 58 | 61 | 64 | 59
mmHg
  Mean @ Baseline | 142.8 [138.7 to 146.9] | 146.8 [142.1 to 151.6] | 143.9 [139.6 to 148.2] | 144.7 [140 to 149.5] | 148 [142.5 to 153.5] | 145.8 [140.4 to 151.1] | 147.4 [142.6 to 152.1] | 149 [143.5 to 154.5]
  Mean of Median SBP @ 12 months: number analyzed (Participants) | 25 | 31 | 25 | 22 | 30 | 31 | 24 | 23
  Mean of Median SBP @ 12 months | 135.1 [127.7 to 142.4] | 136.8 [130.7 to 143] | 138.2 [129.7 to 146.7] | 135.4 [130 to 140.9] | 136.9 [130.5 to 143.2] | 138.8 [131.3 to 146.4] | 139 [131.6 to 146.4] | 138.5 [129.3 to 147.6]
  Mean Change from Baseline: number analyzed (Participants) | 25 | 31 | 25 | 22 | 30 | 31 | 24 | 23
  Mean Change from Baseline | -8.8 [-15 to -2.6] | -8 [-15.3 to -0.7] | -3.2 [-10.1 to 3.7] | -8.8 [-18.1 to 0.5] | -7.3 [-15.6 to 1.1] | -5.4 [-12.3 to 1.6] | -6 [-15.7 to 3.7] | -4.9 [-15.8 to 5.9]

2. Secondary Outcome: Hazard Ratio Analysis of Participant Time From Enrollment Emergency Department Visit to the First PCP Visit
Description: Utilizing multivariable Cox regression analysis, the relationship between mHealth components and attendance at initial Primary Care Physician (PCP) appointment after Emergency Department visit is explored. The analysis adjusts for age, sex, race, presence of a primary care provider, and usage of blood pressure medications. The Hazard Ratio in this context is a measure indicating the relative risk of experiencing the event of interest (time to first PCP visit). A Hazard Ratio greater than 1 implies a greater risk of receipt of a first PCP appointment, and a Hazard Ratio less than 1 implies a lower risk of receipt of a first PCP appointment within 12-month follow-up. The use of Hazard Ratio in this context allows for the assessment of the impact of mHealth components on the timing of primary care engagement while accounting for potential confounding variables. This allows more valuable insights into the effectiveness of these components in facilitating access to primary care visits.
Time Frame: Baseline ED visit (in days)
Population: 211 is all of the participants in each of the eight arms who completed
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- Healthy Behavior Texts: Healthy Behavior Texts: Participants receive daily motivational health behavior texts
- Daily (vs. Weekly) Prompted Self-Measured Blood Pressure: BP Monitoring Daily Via Text Messaging: Daily text messages will prompt participants for BP by home cuff
- Facilitated PCP Appointment Scheduling and Transportation: Physician appointment and transportation scheduling: Participants receive assistance scheduling physician appointment and transportation to those appointments
Arm/Group | Healthy Behavior Texts | Daily (vs. Weekly) Prompted Self-Measured Blood Pressure | Facilitated PCP Appointment Scheduling and Transportation
Number analyzed (Participants) | 211 | 211 | 211
hazard ratio | 0.9 [0.7 to 1.3] | 1.2 [0.9 to 1.6] | 1.2 [0.9 to 1.6]

3. Secondary Outcome: Odds Ratio Analysis of Participants Completing 2 or More Primary Care Visits
Description: Utilizing logistic regression analysis, the probability of participants attending 2 or more primary care visits within a 12-month period is explored. The analysis adjusts for age, sex, race, presence of a primary care provider, and usage of blood pressure medications. The Odds Ratio in this context indicates the likelihood of an event occurring. A higher Odds Ratio suggests an increased likelihood of attending multiple primary care visits, while a lower Odds Ratio indicates a decreased likelihood. The use of Odds Ratio in this context is justified as it allows for the comparison of the likelihood of attending two or more primary care while accounting for covariates. This is useful in logistic regression analysis, where the outcome variable is binary (i.e., attending two or more primary care visits or not) and the focus is on understanding the association between predictor variables and the probability of the outcome.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Healthy Behavior Texts | Daily (vs. Weekly) Prompted Self-Measured Blood Pressure | Facilitated PCP Appointment Scheduling and Transportation
Number analyzed (Participants) | 211 | 211 | 211
Odds Ratio | 0.7 [0.4 to 1.4] | 1.8 [0.9 to 3.6] | 1.7 [0.9 to 3.5]

ADVERSE EVENTS:
Time Frame: 12 months for those who were in the main study; and another 3-6 months for those who opted to continue with the extension study.
Description: Reporting serious adverse events (SAEs) are based on the guidelines of the International Conference on Harmonization (ICH).
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6 | Arm 7 | Arm 8
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/60 | 0/63 | 2/61 | 0/58 | 0/61 | 1/64 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60 | 0/63 | 0/61 | 0/58 | 0/61 | 0/64 | 0/59
Other Adverse Events (participants affected / at risk) | 0/62 | 0/60 | 0/63 | 0/61 | 0/58 | 0/61 | 0/64 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03422718/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03422718/SAP_001.pdf
  • Informed Consent Form (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT03422718/ICF_002.pdf